CLINICAL TRIAL: NCT05010525
Title: A Phase Ib/II Open-label, Multi-centre, Dose Finding Study to Assess the Safety, Pharmacokinetics, and Preliminary Efficacy of ATG 016 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Preliminary Efficacy of ATG 016 Monotherapy in Patients With Advanced Solid Tumors
Acronym: REACH
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on the adjustment of clinical research and development strategy，sponsor decided to terminate the study
Sponsor: Shanghai Antengene Corporation Limited (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG-016-ST-001
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ATG-016-20mg (Experimental): 20 mg QD×5/ week as the initial dose in the Dose Escalation Phase, with a treatment cycle of 21 days,1-5/week will be the initial dose of this study
  Interventions: Drug: ATG-016
- ATG-016-35mg (Experimental): 35 mg QD×5/ week as the initial dose in the Dose Escalation Phase, with a treatment cycle of 21 days,1-5/week will be the initial dose of this study
  Interventions: Drug: ATG-016
- ATG-016-50mg (Experimental): 50 mg QD×5/ week as the initial dose in the Dose Escalation Phase, with a treatment cycle of 21 days,1-5/week will be the initial dose of this study
  Interventions: Drug: ATG-016
- ATG-016-65mg (Experimental): 65 mg QD×5/ week as the initial dose in the Dose Escalation Phase, with a treatment cycle of 21 days,1-5/week will be the initial dose of this study
  Interventions: Drug: ATG-016

INTERVENTIONS:
Drug: ATG-016 — 48 patients enrolled, orally, each 3 week (21-day) a cycle

SUMMARY:
This is A Phase Ib/II Study to Assess the Safety, Pharmacokinetics, and Preliminary Efficacy of ATG 016 Monotherapy in Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is A Phase Ib/II Open-label, Multi-centre, Dose Finding Study to Assess the Safety, Pharmacokinetics, and Preliminary Efficacy of ATG 016 Monotherapy in Patients with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign informed Consent (ICF) prior to any assessment/procedure related to study.
2. Age ≥18 years at ICF signature.
3. Estimated life expectancy of minimum of 12 weeks.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at ICF signature.
5. Subjects must have at least one measurable lesion as defined by RECIST version 1.1.
6. Females of childbearing potential must agree to use effective contraception from the time ICF signature until 180 days after the last dose. Females of childbearing potential include those who are premenopausal and those who are 2 years postmenopausal. Blood pregnancy tests must be negative for female of childbearing potential must have a negative serum pregnancy test at Screening.

Inclusion Criteria Only for Phase Ib study (Dose Escalation and Expansion phase)

1. Histological or cytological confirmation of a solid tumor, and have progressed despite standard therapy(ies), or are intolerant to standard therapy(ies), or have no standard therapy(ies) exists.

Inclusion Criteria Only for Phase II

1. Penile squamous cell carcinomas confirmed by cytology or histology cannot be excised by radical surgery, or postoperative recurrence or metastasis which is not suitable for platinum chemotherapy or platinum resistance or platinum failure.
2. Nasopharyngeal carcinoma

Exclusion Criteria:

Subjects with any of the following conditions will not be enrolled in this study.

1. Central nervous system (CNS) metastases and involvement.
2. A history of bone marrow or organ transplantation.
3. Prior ATG-016 administration or other XPO1 inhibitor treatment.
4. Known to be allergic to the active or inactive ingredients of ATG-016 or drugs with similar chemical structure, or the subject is hypersensitive.
5. Prior therapy with any investigational drugs or systemic anticancer treatment (eg, a period of 5 'half-lives' of drugs, whichever is longer) within 28 days at the time of ICF signature.
6. Received extensive radiation within 28 days at the time of ICF signature or expect to undergo radical radiotherapy during the study period.
7. Received major surgery within 28 days at the time of ICF signature or expect to proceed a major surgical treatment during the study period.
8. Any toxicities unresolved to Grade 1 or baseline from prior anti-tumor therapy (According to NCI-CTCAE 5.0) with the exception of alopecia, within 28 days at the time of ICF signature.
9. Any uncontrolled active infection requiring parenteral treatment of antibiotics, antivirals, or antifungals at the time of ICF signature or within one week of Cycle 1 Day 1 (C1D1). Active hepatitis B virus (HBV) infection (Hepatitis B surface antigen [HBsAg] positive) or active HCV infection (HCV-RNA positive at screening).
10. A history of HIV infection and/or acquired immunodeficiency syndrome.
11. Received immunosuppressive medication within 14 days at the time of ICF signature.
12. Cardiovascular diseases of clinical significance
13. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:
14. Have a history of another primary malignancy within 5 years prior to starting study treatment, with following exceptions: malignancy tumors treated by radical therapy and have not been recurred, such as carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin, papillary thyroid carcinoma, etc.
15. Inability or unwillingness to comply with the requirement for oral drug administration, or presence of a gastrointestinal diseases or other clinical conditions that would compromise the absorption of study drug, eg, refractory nausea and vomiting, inability to swallow the formulated product, or previous significant bowel resection, etc.
16. Active or a history of bleeding within 6 months.
17. Received any live attenuated vaccination within 28 days at the signature of ICF.
18. Judgment by the investigator that the subject should not participate in the study by consideration of the complications or other conditions which might affect their adherence to the protocol.
19. Female subjects who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
MTD in Phase I | 16 months
  MTD will be evaluated using the NCI-CTCAE, Version 5.0
RP2D in Phase I | 16 months
  RP2D will be determined under the guidance of the SRC.
AEs | 25 months
  Toxicity will be graded according to the NCI CTCAE, Version 5.0.
SAEs | 25 months
  Toxicity will be graded according to the NCI CTCAE, Version 5.0.
ORR in Phase II | 25 months
  Based on 2006 IWG Response Criteria, evaluated by IRC: ORR (CR + PR + mCR)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) in Phase I/II | 16 months
  DCR (CR + PR + mCR + HI + SD)
Duration of Response (DOR) in Phase I/II | 12 months
  To evaluate duration of response
Overall Survival (OS） | 12 months
  The estimates of Kaplan-Meier

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, PhD, Principal Investigator — Guoxue lane, Chengdu, Sichuan
Locations (4):
- China (4):
  - The First Affiliated Hospital of Bengbu Medical College Bengbu, Bengbu, Anhui
  - Chongqing Cancer Hospital, Chongqing, Chonqing
  - The First Affiliated Hospital of Xiamen University, Xiaomen, Fujian
  - West China Hospital, Sichuan University, Chengdu, Sichuan